CLINICAL TRIAL: NCT01351857
Title: Multicentre Randomized Controlled Trial of Structured Transition on Diabetes Care Management Compared to Standard Diabetes Care in Adolescents and Young Adults With Type 1 Diabetes
Brief Title: Diabetes Care Management Compared to Standard Diabetes Care in Adolescents and Young Adults With Type 1 Diabetes
Acronym: TransClin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTN1102
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; 17 to 20 years of age
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transition Coordinator (Other): A Transition Coordinator, a Certified Diabetes Educator, will provide transition support and the link between pediatric and adult diabetes care. The Transition Coordinator is central to the intervention and will provide ongoing contact with the medical system as well as education and clinical support where appropriate.
  Interventions: Other: Transition Coordinator
- Current Standard of Care (No Intervention): Subjects in the control group will transition to adult care equal to the intervention group and will differ only by exclusion of Transition Coordinator. Control group will receive the current standard of diabetes care otherwise unchanged. Three months following randomization, subjects in the control group will be referred to the adult endocrinologist in the same way as subjects in the intervention group

INTERVENTIONS:
Other: Transition Coordinator — The Transition Coordinator is central to the intervention and will provide ongoing contact with the medical system as well as education and clinical support where appropriate.
  Arms: Transition Coordinator

SUMMARY:
Structured transition program for adolescents and young adults with Type 1 Diabetes (T1D) improves diabetes clinic attendance as well as glycemic control after transition from pediatric to adult diabetes care.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a structured transition program for adolescents and young adults with Type 1 Diabetes (T1D) improves diabetes clinic attendance and management as well as glycemic control after transition from pediatric to adult diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Established T1D diagnosis for a minimum of one year (chosen to allow time for adjustment to a new diagnosis and more stable disease control).
* Between the ages of 17 and 20 years. It is left to the clinical judgment of the pediatric endocrinologist to determine individually the appropriate age of the transition for each subject
* At least 1 visit during the previous year with the pediatric endocrinologist at a Diabetes Clinic (aim is to minimize the non-adherence with the intervention).
* Ability to participate in all aspects of this clinical trial.
* Written informed consent/assent must be obtained and documented.
* Resident of Ontario.

Exclusion Criteria:

* Pregnant or lactating females or intent to become pregnant during the next 3 years.
* Conditions which in the opinion of the investigator may interfere with the subject's ability to participate in the study.
* Prior enrollment in the current study.
* Current participation in another clinical trial or participation in another clinical trial in the 6 months prior to enrollment.

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2012-04; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who fail to attend at least one outpatient adult endocrinology visit during the second year after transition to adult diabetes care. | 30 months

SECONDARY OUTCOMES:
In the 2 year transfer to adult care-Frequency of A1C (glycated hemoglobin test) | 30 months
  In the 2 year transfer to adult care-Frequency of A1C (glycated hemoglobin test) & mean levels Frequency of retinal exam microalbumin to creatinine ratio fasting lipid profile and foot exam testing Rate of hospitalization/ER visits for acute complications of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Cheril Clarson, MD, Principal Investigator — London Health Sciences Centre - Children's Hospital; Tamara Spaic, Principal Investigator — St. Joseph's Healthcare Centre
Locations (4):
- Canada (4):
  - St. Joseph's Health Care, London, Ontario
  - London Health Sciences Centre - Children's Hospital, London, Ontario
  - Trillium Pediatric Diabetes Clinic, Mississauga, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

REFERENCES:
- [Background] Osgood DW, Foster EM, Courtney ME. Vulnerable populations and the transition to adulthood. Future Child. 2010 Spring;20(1):209-29. doi: 10.1353/foc.0.0047. PMID 20364628
- [Derived] Spaic T, Robinson T, Goldbloom E, Gallego P, Hramiak I, Lawson ML, Malcolm J, Mahon J, Morrison D, Parikh A, Simone A, Stein R, Uvarov A, Clarson C; JDRF Canadian Clinical Trial CCTN1102 Study Group. Closing the Gap: Results of the Multicenter Canadian Randomized Controlled Trial of Structured Transition in Young Adults With Type 1 Diabetes. Diabetes Care. 2019 Jun;42(6):1018-1026. doi: 10.2337/dc18-2187. Epub 2019 Apr 22. PMID 31010873
- [Derived] Spaic T, Mahon JL, Hramiak I, Byers N, Evans K, Robinson T, Lawson ML, Malcolm J, Goldbloom EB, Clarson CL; JDRF Canadian Clinical Trial CCTN1102 Study Group. Multicentre randomized controlled trial of structured transition on diabetes care management compared to standard diabetes care in adolescents and young adults with type 1 diabetes (Transition Trial). BMC Pediatr. 2013 Oct 9;13:163. doi: 10.1186/1471-2431-13-163. PMID 24106787